CLINICAL TRIAL: NCT03816137
Title: An Experimental Medicine Study Modelling the Interaction Between Rationally-designed Synthetic Model Viral Protein Immunogens and the Breadth of the Induced B and T Cell Repertoires.
Brief Title: Modelling the Interaction Between Rationally-designed Synthetic Model Viral Protein Immunogens
Acronym: EAVI2020_01
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: 18HH4893
Record Dates: First submitted 2019-01-22; First posted 2019-01-25 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: HIV-1-infection
Keywords: Antibody; Antibody-dependent cell-mediated cytotoxicity; Neutralizing antibody responses

STUDY DESIGN:
Intervention Model Description: This is a single-blind study with volunteers being randomised into five groups of n=10 (Groups A-E) and eight groups of n=8 (Groups F-M), stratified by gender
Who Masked: Participant, Outcomes Assessor
Masking Description: Volunteers will be blinded to their treatment regimes, and laboratory teams undertaking immunological analysis will be blinded to group and dosing regimen to prevent in-house analysis bias. The clinical team will remain un-blinded throughout.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (13):
- Group A: ConM SOSIP and Mosaic SOSIPs (Active Comparator): ConM SOSIP 100mcg Intramuscular injections into the left or right arm Administered at 0, 3 and 6 months
  Mosaic SOSIPs (Mos3.1 + Mos3.2) 100mcg (2x50mcg) Intramuscular injections into the left or right arm Administered at 12 months only
  Interventions: Biological: ConM SOSIP; Biological: Mosaic SOSIPs
- Group B: EDC ConM SOSIP and Mosaic SOSIPs (Active Comparator): EDC ConM SOSIP 100mcg Intramuscular injections into the left or right arm Administered at 0, 3 and 6 months
  Mosaic SOSIPs (Mos3.1 + Mos3.2) 100mcg (2x50mcg) Intramuscular injections into the left or right arm Administered at 12 months only
  Interventions: Biological: EDC ConM SOSIP; Biological: Mosaic SOSIPs
- Group C: ConS UFO and Mosaic SOSIPs (Active Comparator): ConS UFO 100mcg Intramuscular injections into the left or right arm Administered at 0, 3 and 6 months
  Mosaic SOSIPs (Mos3.1 + Mos3.2) 100mcg (2x50mcg) Intramuscular injections into the left or right arm Administered at 12 months only
  Interventions: Biological: ConS UFO; Biological: Mosaic SOSIPs
- Group D: EDC ConS UFO and Mosaic SOSIPs (Active Comparator): EDC ConS UFO 100mcg Intramuscular injections into the left or right arm Administered at 0, 3 and 6 months
  Mosaic SOSIPs (Mos3.1 + Mos3.2) 100mcg (2x50mcg) Intramuscular injections into the left or right arm Administered at 12 months only
  Interventions: Biological: EDC ConS UFO; Biological: Mosaic SOSIPs
- Group E: ConS UFO and ConM SOSIP and Mosaic SOSIPs (Active Comparator): ConS UFO 100mcg Intramuscular injections into the left or right arm Administered at 0 and 3 months
  ConM SOSIP 100mcg Intramuscular injection into the left or right arm Administered at 6 months
  Mosaic SOSIPs (Mos3.1 + Mos3.2) 100mcg (2x50mcg) Intramuscular injections into the left or right arm Administered at 12 months only
  Interventions: Biological: ConM SOSIP; Biological: ConS UFO; Biological: Mosaic SOSIPs
- Group F: Mosaic SOSIPs and ConM SOSIP and ConS UFO (Active Comparator): Mosaic SOSIP Mos3.1 100mcg Intramuscular injection into the left or right arm Administered at 0 months
  Mosaic SOSIP Mos3.2 100mcg Intramuscular injection into the left or right arm Administered at 2 months
  Mosaic SOSIP Mos3.3 100mcg Intramuscular injection into the left or right arm Administered at 4 months
  ConM SOSIP + ConS UFO 50mcg + 50mcg Intramuscular injections into the left or right arm Administered at 6 months
  Interventions: Biological: ConM SOSIP; Biological: ConS UFO; Biological: Mosaic SOSIPs
- Group G: Mosaic SOSIPs and ConM SOSIP and ConS UFO (Active Comparator): Mosaic SOSIP Mos3.2 100mcg Intramuscular injection into the left or right arm Administered at 0 months
  Mosaic SOSIP Mos3.1 100mcg Intramuscular injection into the left or right arm Administered at 2 months
  Mosaic SOSIP Mos3.3 100mcg Intramuscular injection into the left or right arm Administered at 4 months
  ConM SOSIP + ConS UFO 50mcg + 50mcg Intramuscular injections into the left or right arm Administered at 6 months
  Interventions: Biological: ConM SOSIP; Biological: ConS UFO; Biological: Mosaic SOSIPs
- Group H: Mosaic SOSIPs and ConM SOSIP and ConS UFO (Active Comparator): Mosaic SOSIP Mos3.3 100mcg Intramuscular injection into the left or right arm Administered at 0 months
  Mosaic SOSIP Mos3.2 100mcg Intramuscular injection into the left or right arm Administered at 2 months
  Mosaic SOSIP Mos3.1 100mcg Intramuscular injection into the left or right arm Administered at 4 months
  ConM SOSIP + ConS UFO 50mcg + 50mcg Intramuscular injections into the left or right arm Administered at 6 months
  Interventions: Biological: ConM SOSIP; Biological: ConS UFO; Biological: Mosaic SOSIPs
- Group I: Mosaic SOSIPs and ConM SOSIP and ConS UFO (Active Comparator): Mosaic SOSIPs (Mos3.1 + Mos3.2 + Mos3.3) 100mcg (3x33mcg) Intramuscular injections into the left or right arm Administered at 0, 2 and 4 months
  ConM SOSIP + ConS UFO 50mcg + 50mcg Intramuscular injections into the left or right arm Administered at 6 months
  Interventions: Biological: ConM SOSIP; Biological: ConS UFO; Biological: Mosaic SOSIPs
- Group J: 763 SOSIP (Active Comparator): 763 SOSIP 100mcg Intramuscular injections into the left or right arm Administered at 0, 2 and 4 months
  Interventions: Biological: 763 SOSIP
- Group K: AMC011 SOSIP (Active Comparator): AMC011 100mcg Intramuscular injections into the left or right arm Administered at 0, 2 and 4 months
  Interventions: Biological: AMC011 SOSIP
- Group L: 763 SOSIP and AMC011 SOSIP (Active Comparator): 763 SOSIP and AMC011 50mcg + 50mcg Intramuscular injections into the left or right arm Administered at 0, 2 and 4 months
  Interventions: Biological: 763 SOSIP; Biological: AMC011 SOSIP
- Group M: 763 SOSIP and AMC011 SOSIP and ConM SOSIP and Mosaic SOSIPs (Active Comparator): 763 SOSIP and AMC011 SOSIP and ConM SOSIP and Mos3.1 and Mos3.2 SOSIPs each at 20mcg Intramuscular injections into the left or right arm Administered at 0, 2 and 4 months
  Interventions: Biological: ConM SOSIP; Biological: Mosaic SOSIPs; Biological: 763 SOSIP; Biological: AMC011 SOSIP

INTERVENTIONS:
Biological: ConM SOSIP — Recombinant HIV-1 trimeric gp140 Env protein: ConM SOSIP gp140. Model immunogens will be used at the dosage of 20 mcg or 50 mcg or 100 mcg and will be admixed with 500 mcg MPLA formulated in liposomes and administered by intramuscular injection into the left or right deltoid muscle.
  Arms: Group A: ConM SOSIP and Mosaic SOSIPs; Group E: ConS UFO and ConM SOSIP and Mosaic SOSIPs; Group F: Mosaic SOSIPs and ConM SOSIP and ConS UFO; Group G: Mosaic SOSIPs and ConM SOSIP and ConS UFO; Group H: Mosaic SOSIPs and ConM SOSIP and ConS UFO; Group I: Mosaic SOSIPs and ConM SOSIP and ConS UFO; Group M: 763 SOSIP and AMC011 SOSIP and ConM SOSIP and Mosaic SOSIPs
Biological: EDC ConM SOSIP — Chemically fixed version of recombinant HIV-1 trimeric gp140 Env: EDC ConM SOSIP. Model immunogens will be used at the dosage of 100 mcg and will be admixed with 500 mcg MPLA formulated in liposomes and administered by intramuscular injection into the left or right deltoid muscle.
  Arms: Group B: EDC ConM SOSIP and Mosaic SOSIPs
Biological: ConS UFO — Recombinant HIV-1 trimeric gp140 Env protein: ConS UFO gp140. Model immunogens will be used at the dosage of 50 mcg or 100 mcg and will be admixed with 500 mcg MPLA formulated in liposomes and administered by intramuscular injection into the left or right deltoid muscle
  Arms: Group C: ConS UFO and Mosaic SOSIPs; Group E: ConS UFO and ConM SOSIP and Mosaic SOSIPs; Group F: Mosaic SOSIPs and ConM SOSIP and ConS UFO; Group G: Mosaic SOSIPs and ConM SOSIP and ConS UFO; Group H: Mosaic SOSIPs and ConM SOSIP and ConS UFO; Group I: Mosaic SOSIPs and ConM SOSIP and ConS UFO
Biological: EDC ConS UFO — Chemically fixed version of recombinant HIV-1 trimeric gp140 Env : EDC-ConS UFO. Model immunogens will be used at the dosage of 100 mcg and will be admixed with 500 mcg MPLA formulated in liposomes and administered by intramuscular injection into the left or right deltoid muscle.
  Arms: Group D: EDC ConS UFO and Mosaic SOSIPs
Biological: Mosaic SOSIPs — Mosaic gp140 Env trimers (Mos3.1, Mos3.2, Mos3.3) designed to overcome the immunodominance of hypervariable regions of Env. The immunogen will be used at the dosage of 100 mcg (100mcg or 2 x 50 mcg or 3 x 33 mcg) or at 40 mcg (2 x 20mcg) and will be admixed with 500 mcg MPLA formulated in liposomes and administered by intramuscular injection into the left or right deltoid muscle.
  Arms: Group A: ConM SOSIP and Mosaic SOSIPs; Group B: EDC ConM SOSIP and Mosaic SOSIPs; Group C: ConS UFO and Mosaic SOSIPs; Group D: EDC ConS UFO and Mosaic SOSIPs; Group E: ConS UFO and ConM SOSIP and Mosaic SOSIPs; Group F: Mosaic SOSIPs and ConM SOSIP and ConS UFO; Group G: Mosaic SOSIPs and ConM SOSIP and ConS UFO; Group H: Mosaic SOSIPs and ConM SOSIP and ConS UFO; Group I: Mosaic SOSIPs and ConM SOSIP and ConS UFO; Group M: 763 SOSIP and AMC011 SOSIP and ConM SOSIP and Mosaic SOSIPs
Biological: 763 SOSIP — HIV-1 envelope sequence, identified from two HIV infected individuals that displayed HIV neutralisation breadth early in infection (less than 12 months). The immunogen will be used at the dosage of 20 mcg or 50mcg or 100mcg and will be admixed with 500 mcg MPLA formulated in liposomes and administered by intramuscular injection into the left or right deltoid muscle.
  Arms: Group J: 763 SOSIP; Group L: 763 SOSIP and AMC011 SOSIP; Group M: 763 SOSIP and AMC011 SOSIP and ConM SOSIP and Mosaic SOSIPs
Biological: AMC011 SOSIP — HIV-1 envelope sequence, identified from two HIV infected individuals that displayed HIV neutralisation breadth early in infection (less than 12 months). The immunogen will be used at the dosage of 20 mcg or 50mcg or 100mcg and will be admixed with 500 mcg MPLA formulated in liposomes and administered by intramuscular injection into the left or right deltoid muscle.
  Arms: Group K: AMC011 SOSIP; Group L: 763 SOSIP and AMC011 SOSIP; Group M: 763 SOSIP and AMC011 SOSIP and ConM SOSIP and Mosaic SOSIPs

SUMMARY:
The objective of this experimental medicine study is to determine the extent to which different prime-boost combinations influence serum neutralising antibody breadth and associated B and T cells responses.

The investigators hypothesise that the different prime-boost model immunogen combinations will have differential impact on: the magnitude and breadth of induced serum neutralising antibodies; and the induced B- and T-cell responses in peripheral blood.

The investigators will investigate this by challenging the immune system of healthy adults with various model immunogens based on HIV-1 Env (ConM and ConS, with and without EDC stabilisation; Mos3.1, Mos3.2 and Mos3.3, and AMC011 and 763 SOSIP) in different prime-boost combinations.

DETAILED DESCRIPTION:
One of the most effective arms of the human immune system is the ability of very low concentrations of antibody proteins to bind to viruses, bacteria and toxins and "neutralise" their activity or ability to infect. In contrast to cellular immunity, which may cause tissue destruction and pathology, antibody-mediated immunity can be very passive, while completely preventing infection. How antibodies bind their targets varies enormously, ranging from unhelpful "blocking" antibodies or narrowly focussed neutralising antibodies, to highly protective "broadly neutralising" antibodies (bNAbs) that can neutralise a wide range of strains of the same pathogen. Such bNAbs are especially sought after in virus infections such as HIV, influenza and others where the virus mutates to evade immune responses that are too narrow or focussed. Antibodies arise when an "immunogen" (an immunogen is anything that induces an immune response, typically a foreign protein) is taken up by the immune system and shown to white blood cells - T and B cells - by specialised immune cells. In some cases the T and B cells bind the immunogens to receptors on their surface, triggering an immune response in which T cells "help" B cells to manufacture specific antibodies. The events around how the protein is processed into manageable pieces, shown to the T and B cells, and the pattern of chemical signals produced by the immune cells is highly complex, but eventually determines how broad the antibody response will be (its breadth). For infections like HIV and influenza, decades of research and clinical vaccine trials have had limited or no success. To take HIV as an example, investigators have an almost complete lack of understanding of how immunogens interact with the naive human B cell receptor (BCR) repertoire and the pathways required to induce bNAbs during an infection or after an immunisation. Animal models have failed as the naïve, germline encoded, B cell antibody receptor repertoires of non-human species are sufficiently different from those of humans to render design and selection of vaccine based on non-human species problematic. Additionally, bNAbs isolated from HIV-1-infected individuals have structural features that occur rarely or not at all in other mammals, such as unusually long loop-binding regions (CDRH3 loops) required to penetrate past glycans on the surface of the envelope spike that shield key neutralising epitopes. There is therefore a critical need to better understand, in human experimental medicine models of immune challenge, how immunogens and B/T cells interact in the development of protective bNAb anti-viral responses.

The approach by the investigators to resolving this impasse is to challenge the human immune system with rationally-designed model immunogens to determine the structural and other characteristics required to drive human B cell antibody responses towards neutralisation breadth. The investigators have selected HIV as an experimental model as there is a reasonable understanding about the specificity and function of anti-HIV bNAbs, as well as an urgent need to identify novel immunisation approaches following decades of failed or poorly successful trials. There is also a huge database of safety using HIV proteins as immunogens, and the technological expertise to design and manufacture HIV viral proteins. Assays for HIV neutralising activity are also well established in the study team's laboratories. Although focussed on HIV, the investigators' findings will be applicable to other viral infections.

The model immunogens proposed in the experimental medicine studies are unlikely to be suitable as vaccines, and any clinical development would require iterative cycles of design refinement and development based on immunological insights gleaned from these experimental investigations. Therefore, the focus is on in-depth characterisation of the elicited immune response to rationally-designed model immunogens that may inform the design process of actual vaccines. This experimental medicine approach is only now possible due to unprecedented progress in abilities to study the human immune system and to obtain complete information on immune responses to vaccination, since performing research on the human immune system is now almost as easy as it has been in mice. The main focus of this study will be to determine which of the design strategies is able to prime human germline (naive) B cells and drive antibody responses towards induction of neutralising antibody breadth.

The investigators' range of model immunogens will be based on the envelope (Env) glycoprotein of HIV-1, which is the only target of neutralising antibodies, and therefore the only virally-encoded immunogen relevant for induction of such antibodies by immunisation. To ensure reproducibility of results and the highest level of volunteer safety, all immunogens will be manufactured under cGMP, using techniques applied to vaccine immunogens.

Env has extensive amino acid variation, structural and conformational instability, and immunodominance of hypervariable regions. The study team designed soluble immunogens that closely mimic the native viral trimer in situ, but that incorporate design strategies that may alter the intrinsic viral immune evasion mechanisms. Env is made up of three identical complexes (trimers) each of which contains two molecules, gp120 and gp41 that can be modified to make a soluble molecule called gp140, upon which the investigators' immunogens are based. Investigators have developed model consensus gp140 Env trimers (consensus of all global strains) designed to prime B cell responses to common epitopes represented in all HIV-1 subtypes. Investigators have utilised two design strategies to stabilise these in a native-like conformation: ConM SOSIP and ConS UFO.

The ConM SOSIP trimer includes novel mutations that include the incorporation of a disulphide linkage between the gp120 and gp41 ectodomain (making up gp140) which prevents their disassociation into monomer subunits. The ConS UFO includes a short flexible amino-acid linker to tether the gp120 and gp41 subunits together as an alternative strategy to prevent dissociation of the Env trimer. The investigators wish to test both designs to determine the effect on B cell repertoire. To further stabilize global architecture, the investigators employed an EDC crosslinking approach that has been shown to conserve bNAb epitopes, reduce non-antiviral antibody responses, and enhance overall immunogen stability. Thus, in Part 1 of this study the investigators will test EDC ConM SOSIP and EDC ConS UFO versions in parallel.

A critical adjunct to the investigators' consensus-based model design is to use a cocktail of three mosaic gp140 Env trimers as a boost (Part 2) to overcome the immunodominance of hypervariable regions of Env and to determine whether this will focus antibody responses towards conserved neutralisation epitopes. While designed using computer algorithms, these mosaics represent authentic Env structures that are fully functional and native in their conformation. The investigators' novel designs aim to eliminate unwanted immunodominant antibody responses and focus B cells towards highly conserved supersites of vulnerability on Env, with particular emphasis on quaternary bNAb epitopes. The extent to which these different strategies may induce neutralising breadth, and the identification of the mechanisms and drivers involved, can only be determined empirically through human immunogen challenge studies.

Two HIV-1 envelope sequences (AMC011 SOSIP and 763 SOSIP) will also be used as immunogens in some of the study groups. The EAVI2020 programme has found these to be associated with the early induction of broadly neutralising antibodies. The sequences were identified from two HIV infected individuals who displayed HIV neutralisation breadth early in infection (less than 12 months). This is unusual as typically neutralisation breadth is only seen to develop in < 5% of subjects and only after a period of more than 2 years. The investigators seek to test the hypothesis that these two envelope sequences may display unique potential to prime and/or drive the induction of broadly neutralising antibody responses in HIV negative healthy volunteers. To test this hypthesis the EAVI2020 consortium has manufactured stabilised versions of these two envelope proteins to GMP. These will be used alone and in various combinations with consensus and mosaic immunogens to determine the extent to which they can drive the induction of broadly neutralising antibodies. Responses to these unique envelope sequences will be compared and contrasted to the consensus and mosaic immunogens evaluated in other study groups.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female volunteers aged between 18 and 55 years.
2. Available for ALL follow-up visits for the duration of the study.
3. Entered and clearance obtained from The Over volunteering Prevention System (TOPS) database (to avoid impact of any co-administered investigational products or treatments on our outcomes).
4. Women of childbearing potential willing to use a highly effective method of contraception for the duration of the study until a minimum of 12 weeks after the final injection. Periodic abstinence (calendar, symptothermal and post-ovulation methods) and withdrawal are not acceptable methods of contraception.
5. Willing and able to give written informed consent.

Exclusion Criteria:

1. History of any medical, psychological or other condition, clinically significant laboratory result at screening, or use of any medications which, in the opinion of the investigators, would interfere with the study objectives or volunteers safety.
2. Any history of angioedema.
3. History of urticaria deemed significant by the Chief Investigator.
4. HIV-1 or HIV-2 antibody positive or indeterminate upon screening, or history of receipt of Env-based HIV immunogens (which would render the volunteers non-naive to the model immunogens).
5. Unable to read and/or speak English to a fluency level adequate for the full comprehension of study procedures and consent.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 117 (Actual)
Dates: Start 2019-03-19 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Neutralising antibodies to virus expressing ConM and ConS envelopes | 6 Months
  Serum titres of neutralising antibodies to virus expressing ConM and ConS envelopes
Neutralising antibodies to virus expressing Mosaic envelopes | 12 Months
  Serum titres of neutralising antibodies to virus expressing Mosaic envelopes (Mos3.1, Mos3.2, Mos3.3)
Neutralising antibodies to virus expressing AMC011 and 763 SOSIP envelopes | 4 months
  Serum titres of neutralising antibodies to virus expressing AMC011 and 763 SOSIP envelopes

CONTACTS AND LOCATIONS:
Overall Officials: Katrina Pollock, Principal Investigator — Imperial College London
Locations (1):
- NIHR Imperial Clinical Resarch Facility, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Results from this study will be disseminated locally and to the wider scientific community at conferences and in published open-access peer-reviewed journals, as appropriate. Any data used for publication will be fully anonymised. The investigators plan to publish the data and hold onto the data for 10 years.
Supporting Information: CSR
Time Frame: 12 months from when the experimental study officially closes
Access Criteria: Directly from Professor Robin Shattock (r.shattock@imperial.ac.uk)

REFERENCES:
- [Derived] Pollock KM, Cheeseman HM, McFarlane LR, Day S, Tolazzi M, Turner HL, Joypooranachandran J, Shramko K, Dispinseri S, Mundsperger P, Bontjer I, Lemm NM, Coelho S, Tanaka M, Cole T, Korber B, Katinger D, Sattentau QJ, Ward AB, Scarlatti G, Sanders RW, Shattock RJ. Experimental medicine study with stabilised native-like HIV-1 Env immunogens drives long-term antibody responses, but lacks neutralising breadth. EBioMedicine. 2025 Feb;112:105544. doi: 10.1016/j.ebiom.2024.105544. Epub 2025 Jan 2. PMID 39753033

DOCUMENTS (2):
  • Study Protocol (2022-11-14): https://cdn.clinicaltrials.gov/large-docs/37/NCT03816137/Prot_000.pdf
  • Informed Consent Form (2022-01-25): https://cdn.clinicaltrials.gov/large-docs/37/NCT03816137/ICF_001.pdf